CLINICAL TRIAL: NCT04691063
Title: A Multi-center, Randomized, Double-blinded, Phase III Trial of SHR-1316 or Placebo in Combination With Chemo-radiotherapy in Patients With Limited-stage Small-cell Lung Cancer.
Brief Title: The Study is Being Conducted to Evaluate the Efficacy and Safety of SHR-1316 in Combination With Chemo-radiotherapy in Patients With LS-SCLC.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1316-III-302
Record Dates: First submitted 2020-12-25; First posted 2020-12-31 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2020-12

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin

STUDY DESIGN:
Intervention Model Description: SHR-1316 in combination with chemo-radiotherapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-1316; Carboplatin; Etoposide；Radiotherapy
- Treatment group B (Placebo Comparator)
  Interventions: Drug: Palcebo; Carboplatin; Etoposide；Radiotherapy

INTERVENTIONS:
Drug: SHR-1316; Carboplatin; Etoposide；Radiotherapy — SHR-1316; Carboplatin; Etoposide；Radiotherapy（Part 1 and Part 2）
  Arms: Treatment group A
Drug: Palcebo; Carboplatin; Etoposide；Radiotherapy — Palcebo; Carboplatin; Etoposide；Radiotherapy（Part 2）
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR-1316 in combination with chemo-radiotherapy in patients with LS-SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-75 years of age.
2. Subjects with histologically confirmed Limited-Stage SCLC without previous systematic treatment.
3. ECOG PS 0~1.
4. At least 1 measurable lesion as defined by RECIST v1.1.
5. Adequate organ function.
6. Female subjects of childbearing potential or male subjects must be willing to use a recognized effective contraceptive measure during the study and within 3 months after the last dose of the study drug. And female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose.
7. Signed the informed consent form.

Exclusion Criteria:

1. Mixed SCLC or NSCLC.
2. Subjects who previously received systemic antitumor or Immune checkpoint inhibitor therapy.
3. Extensive-stage SCLC.
4. Subjects who is surgically resectable.
5. Subjects with malignant pleural effusion.
6. Subjects highly suspected of interstitial lung disease, or with conditions that may interfere with the testing or management of suspected treatment-related pulmonary toxicities, or other moderate to severe diseases that seriously affect pulmonary function.
7. Active, known, or suspected autoimmune diseases.
8. History of malignant tumors.
9. Subjects with severe cardiovascular disease.
10. Events of arterial/venous thrombosis within 6 months prior to the first dose.
11. Subjects with serious infection.
12. Subjects with active pulmonary tuberculosis (TB).
13. Subjects with immunodeficiency diseases.
14. Subjects with active hepatitis B virus or hepatitis C virus infection.
15. Systemic immunosuppressants administation within 14 days prior to the first dose.
16. Subjects who received major surgery within 28 days prior to the first dose.
17. Subjects who plan to receive or have received live vaccines within 28 days prior to the first dose.
18. Subjects who have previously received tissue/organ transplants.
19. Subjects with history of severe allergic reactions to monoclonal antibodies/fusion protein drugs.
20. Subjects with mental illness, alcohol abuse, inability to quit smoking, and drug or substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
OS | up to 36 months
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China